CLINICAL TRIAL: NCT07009821
Title: SCREENING EmoCamp_ Analysis of Major Haemoglobinopathies Among Newborns in the Campania Region
Brief Title: Neonatal Screening for Haemoglobinopathies EmoCamp
Acronym: EmoCamp
Status: Not yet recruiting | Type: Observational
Sponsor: Maddalena Casale (Other)
Responsible Party: Sponsor-Investigator, Maddalena Casale, Associate Professor in Pediatrics, University of Campania Luigi Vanvitelli
Organization: University of Campania Luigi Vanvitelli (Other)
Other Study IDs: EmoCamp
Record Dates: First submitted 2025-05-28; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: SCD
Keywords: SCD; neonatal screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hereditary haemoglobin defects defined under the term haemoglobinopathies represent the most frequent congenital diseases worldwide.

The proposed observational study is aimed at determining the prevalence of haemoglobinopathies in newborns in the Campania Region. The neonatal screening test will be performed at the birth centers in Campania Region, before the newborn's discharge, at the same time as the sampling for neonatal screening required by law.

The main objective of this study is to evaluate the feasibility and impact of the screening programme performed at the birth centers on the earliness of diagnosis and the annual rate of sickle cell anaemia diagnosis in children. The secondary objective is to evaluate the benefits of early diagnosis of SCD in children as measured by two endpoints:

* Improved disease management and early initiation of conventional therapy with reduction of complications, potentially fatal;
* Difference between costs related to the neonatal screening programme and estimated costs related to conventional screening and treatment resulting from complications that may arise with late diagnosis.

DETAILED DESCRIPTION:
In the first years of life, unrecognised and untreated SCD patients have a high risk of mortality caused mainly by infection, splenic sequestration and stroke; the mortality risk is 1.1% per year in the first 10 years, but peaks in the first 3 years.

Screening may be universal or targeted, involving the neonatal population only or different age groups. Early diagnosis of disease and subsequent patient care, with timely initiation of antibiotic prophylaxis, vaccinations and parental education to recognise symptoms or signs of risk, has been shown to be effective in drastically reducing morbidity and mortality.

In Italy, newborns are screened at birth and this occasion therefore appears to be the most suitable time to perform the rapid test for the diagnosis of haemoglobinopathies.

The required amount of sample, taken from the newborn's heel, corresponds to 2 drops of blood. Subsequently, the blood sample will be blotted onto a special card made of bibula paper and absorbed by it.

The card, duly retained by the birth centers, will be sent to the Molecular and Cellular Biology laboratory of the Department of Women, Children and General and Specialist Surgery AOU-- Università degli Studi della Campania 'Luigi Vanvitelli' where the screening test will be performed.

In the event of a negative screening test, parents or legal guardians will not be recalled from the centre.

In the event of a positive screening test, parents or legal guardians will be called back by the U.O. Paediatric Haematology and Oncology centre of the AOU Luigi Vanvitelli in Naples to continue the diagnostic procedure and the taking into care of the affected subject, according to clinical practice: prescription blood count+ sideremia+ transferrin+ ferritin+ HPLC+ globin genes study.

Specifically, the test detects normal haemoglobins (F and A) and the most common haemoglobin variants: S, D, C and E.

The screening test makes it possible to anticipate a diagnosis that is often made in emergency situations, sometimes very serious or fatal, and at the same time represents a saving of NHS and SNR resources.

ELIGIBILITY:
Inclusion Criteria:

* newborns at higher risk of disease.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The test will be carried out on all newborns in the Campania region after signing the specific informed consent of their parents or legal guardians.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
determination of haemoglobin fractions | Perioperative/Periprocedural
  Patients were assessed for the presence of abnormal haemoglobin fractions by means of the HPLC method on a peripheral blood drop

CONTACTS AND LOCATIONS:
Overall Officials: Maddalena Casale, Professor, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Azienda Ospedaliera Universitaria "Luigi Vanvitelli", Napoli, Italy, Italy

REFERENCES:
- [Background] Associazione Italiana Ematologia Oncologia Pediatrica. Raccomandazioni per il trattamento della Drepanocitosi in Italia. 2018.
- [Background] Colombatti R, Martella M, Cattaneo L, Viola G, Cappellari A, Bergamo C, Azzena S, Schiavon S, Baraldi E, Dalla Barba B, Trafojer U, Corti P, Uggeri M, Tagliabue PE, Zorloni C, Bracchi M, Biondi A, Basso G, Masera N, Sainati L. Results of a multicenter universal newborn screening program for sickle cell disease in Italy: A call to action. Pediatr Blood Cancer. 2019 May;66(5):e27657. doi: 10.1002/pbc.27657. Epub 2019 Feb 5. PMID 30724025
- [Background] Desselas E, Thuret I, Kaguelidou F, Benkerrou M, de Montalembert M, Odievre MH, Lesprit E, Rumpler E, Fontanet A, Pondarre C, Brousse V. Mortality in children with sickle cell disease in mainland France from 2000 to 2015. Haematologica. 2020 Sep 1;105(9):e440-443. doi: 10.3324/haematol.2019.237602. No abstract available. PMID 33054059
- [Background] Serjeant GR, Chin N, Asnani MR, Serjeant BE, Mason KP, Hambleton IR, Knight-Madden JM. Causes of death and early life determinants of survival in homozygous sickle cell disease: The Jamaican cohort study from birth. PLoS One. 2018 Mar 1;13(3):e0192710. doi: 10.1371/journal.pone.0192710. eCollection 2018. PMID 29494636
- [Background] Shet AS, Lizarralde-Iragorri MA, Naik RP. The molecular basis for the prothrombotic state in sickle cell disease. Haematologica. 2020 Oct 1;105(10):2368-2379. doi: 10.3324/haematol.2019.239350. PMID 33054077
- [Background] Casale M, Scianguetta S, Palma T, Pinfildi L, Vallefuoco G, Capellupo MC, Roberti D, Perrotta S. Screening for sickle cell disease by point-of-care tests in Italy: pilot study on 1000 at risk children. Eur J Pediatr. 2025 Jan 28;184(2):157. doi: 10.1007/s00431-025-05988-y. PMID 39875760
- [Background] National Institutes of Health National Heart, Lung, and Blood Institute. Division of Blood Diseases and Resources. The Management of Sickle Cell Disease. NIH PUBLICATION NO. 02-2117. 2008.
- [Background] McGann PT, Schaefer BA, Paniagua M, Howard TA, Ware RE. Characteristics of a rapid, point-of-care lateral flow immunoassay for the diagnosis of sickle cell disease. Am J Hematol. 2016 Feb;91(2):205-10. doi: 10.1002/ajh.24232. Epub 2015 Nov 26. PMID 26537622
- [Background] Kanter J, Telen MJ, Hoppe C, Roberts CL, Kim JS, Yang X. Validation of a novel point of care testing device for sickle cell disease. BMC Med. 2015 Sep 16;13:225. doi: 10.1186/s12916-015-0473-6. PMID 26377572
- [Background] Darbari DS, Sheehan VA, Ballas SK. The vaso-occlusive pain crisis in sickle cell disease: Definition, pathophysiology, and management. Eur J Haematol. 2020 Sep;105(3):237-246. doi: 10.1111/ejh.13430. Epub 2020 May 19. PMID 32301178